CLINICAL TRIAL: NCT06716138
Title: A Phase 1 Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of ANS03 as a Single Agent in Participants With Locally Advanced or Metastatic Solid Tumors Harboring a ROS1 or NTRK Alteration
Brief Title: A Study to Investigate ANS03 in Participants With Locally Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Avistone Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANS03-I-01
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Locally Advanced or Metastatic Solid Tumors Harboring a ROS1 or NTRK Alteration
Keywords: ROS1/NTRK; ANS03

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ANS03 monotherapy (Experimental)
  Interventions: Drug: ANS03

INTERVENTIONS:
Drug: ANS03 — ANS03 is a rationally next generation TKI targeting both ROS1 and NTRK developed by Shenzhen Avistone Biotechnology (the sponsor).

SUMMARY:
This is a first-in-human Phase I, multi-center, open-label study of ANS03 in patients with advanced solid tumors. The study evaluates the safety, tolerability, preliminary efficay, pharmacokinetics, anti-tumor activity of ANS03 as monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status: 0-2
* Life expectancy ≥ 12 weeks
* Measurable disease per RECIST v1.1
* Adequate organ and marrow function as defined in the protocol
* With documentation of ROS1 or NTRK alteration

Exclusion Criteria:

* Active infection including tuberculosis and HBV, HCV or HIV
* Known active or untreated CNS metastases
* Participants with carcinomatous meningitis or meningeal metastases, or spinal cord compression
* Participants with serious cardiovascular or cerebrovascular diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | From the time of first dose to 28 days post last dose of ANS03
  Number of patients with adverse events by system organ class and preferred term
Incidence of Serious Adverse Events (SAEs) | From time of first dose to 28 days post last dose of ANS03
  Number of patients with serious adverse events by system organ class and preferred term
Incidence of dose-limiting toxicities (DLT) as defined in the protocol | From time of first dose of ANS03 to end of DLT period (approximately 30 days)
  Number of patients with at least 1 dose-limiting toxicity (DLT), which is any toxicity defined as a DLT in the Clinical Study Protocol
Incidence of baseline laboratory finding, ECG and vital signs changes | From time of first dose to 28 days post last dose of ANS03
  measured by laboratory and vital sign variables over time including change from baseline
Proportion of patients with radiological response (ORR) | From date of first dose of ANS03 until progression, or the last evaluable assessment in the absence of progression （approximately 2 years)
  Assessed by overall response rate (ORR) defined as the proportion of patients who have a confirmed complete or partial radiological response by the Investigator according to RECIST v1.1

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From date of first dose of ANS03 up until progression, or the last evaluable assessment in the absence of progression (approximately 2 years)
  The percentage or number of patients with a confirmed investigator assessed complete or partial response according to response criteria in solid tumours (RECIST v1.1)
Duration of Response (DoR) | From date of first dose of ANS03 up until progression, or the last evaluable assessment in the absence of progression (approximately 2 years)
  The time from date of first response until date of disease progression or last evaluable assessment (RECIST v1.1) in the absence of progression
Disease Control Rate (DCR) | From date of first dose of ANS03 up until progression, or the last evaluable assessment in the absence of progression (approximately 2 years)
  The percentage of patients with confirmed CR or PR or having SD maintained (RECIST v1.1)
Progression free Survival (PFS) | From date of first dose of ANS03 up until date of progression or death due to any cause (approximately 2 years)]
  The time from first dose until RECIST 1.1 defined disease progression or death due to any cause
Overall Survival (OS) | From date of first dose of ANS03 up until the date of death due to any cause (approximately 2 years)
  The time from the date of the first dose of study treatment until death due to any cause
Pharmacokinetics of ANS03: Plasma PK concentrations | From date of first dose up until 28 days post last dose
  Measurement of plasma concentrations of ANS03, total antibody and total unconjugated warhead
Pharmacokinetics of ANS03: Area under the concentration time curve (AUC) | From date of first dose up until 28 days post last dose
  Measurement of PK parameters: Area under the concentration time curve (AUC)
Pharmacokinetics of ANS03: Maximum plasma concentration of the study drug (C-max) | From date of first dose up until 28 days post last dose
  Measurement of PK parameters: Maximum observed plasma concentration of the study drug (C-max)
Pharmacokinetics of ANS03: Time to maximum plasma concentration of the study drug (T-max) | Frame: From date of first dose up until 28 days post last dose
  Measurement of PK parameters: Time to maximum observed plasma concentration of the study drug (T-max)
Pharmacokinetics of ANS03: Clearance | From date of first dose up until 28 days post last dose
  Measurement of PK parameters: the volume of plasma from which the study drug is completely removed per unit time (Clearance)
Pharmacokinetics of ANS03: Half-life | From date of first dose up until 28 days post last dose
  Measurement of PK parameters: Terminal elimination half-life (t 1/2)

CONTACTS AND LOCATIONS:
Locations (5):
- Research Site, New York, New York, United States
- China (4):
  - Research Site, Fuzhou, Fujian
  - Research Site, Guangzhou, Guangdong
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Chengdu, Sichuan